CLINICAL TRIAL: NCT04716517
Title: Clinical Evaluation of Bulk-fill Alkasite Restoration Versus Resin Modified Glass Ionomer in Adult Patients With Class V Carious Lesions Over One Year Period: Randomized Clinical Trial
Brief Title: Clinical Evaluation of Bulk-fill Alkasite Restoration Versus Resin Modified Glass Ionomer in Adult With Class V Carious
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hadeel alsalamony, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 381020
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cervical Lesion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cention N (Experimental): Intervention Alkasite Restoration will be used to restore cervical carious in adult patients.
  Interventions: Other: Alkasite bioactive restorative material.
- Resin Modified Glass Ionomer (Active Comparator): Comparator Resin-modified glass ionomer material will be used to restore cervical carious in adult patients.
  Interventions: Other: Resin Modified Glass Ionomer

INTERVENTIONS:
Other: Alkasite bioactive restorative material. — Alkasite restorative is a category of filling material, like compomer, and is essentially a subgroup
  of the composite resin. Cention N is a urethane dimethacrylate (UDMA)-based, self-curing powder/liquid restorative with optional additional light curing. The liquid comprises of dimethacrylates and initiators, while the powder contains various glass fillers, initiators, and pigments. It is radio opaque and contains alkaline glass fillers capable of releasing fluoride, calcium, and hydroxide ions. Due to the sole use of cross-linking methacrylate monomers in combination with a stable, efficient self-cure initiator, Cention N displays a high polymer network density and degree of polymerization over the complete depth of the restoration.
  Other Names: (Cention N).
  Arms: Cention N
Other: Resin Modified Glass Ionomer — The resin-modified glass ionomer materials are hybrid materials of traditional glass ionomer cement with a small addition of light-curing resin, and hence exhibit properties intermediate to the two, with some characteristics superior to conventional glass ionomer materials
  Arms: Resin Modified Glass Ionomer

SUMMARY:
Cention N will have the same clinical performance as resin-modified glass ionomer in cervical carious lesions. Evaluation of restorations will be done at baseline, six months, and one year according (USPHS) criteria.

DETAILED DESCRIPTION:
In this study, Class V carious lesions were restored using two different restorative materials either resin modified glass ionomer or Cention N restorative materials. This study will be held in the restorative clinic at Future University in Egypt. Patients will be assessed for medical and dental histories first. Then an examination of the patients will be done using visual inspection by using a dental mirror and probe. Eligible patients according to inclusion and exclusion criteria will be informed about all procedures with follow up time if they accept, 12 their signature on written informed consents will be obtained. Eligible participants will be randomly divided into two groups according to the type of restoration they will be received. The first group (A) will be received resin modified glass ionomer restorative material and the second group (B) will be received Cention N restorative materials. Each restoration will be evaluated for clinical parameters after finishing and polishing at baseline and regular recalls of 6 months and one year.

The restorations will be clinically examined according to modified USPHS criteria in terms of marginal adaptation, anatomic form, color match, marginal discoloration, secondary caries, postoperative sensitivity and retention. The information that will be obtained will be collected and statistically analyzed

ELIGIBILITY:
Inclusion criteria:

* Patients with High caries risk.
* Patients with poor oral hygiene.
* Patients with untreated cervical caries lesion.
* patient aging ≥18 years.
* Absence of tooth mobility
* Absence of abnormal occlusion.
* Patients with good likelihood of recall availability.

Exclusion criteria:

* Patients with cervical caries lesions need crown restoration.
* Non-vital teeth.
* Evidence of parafunctional habits.
* Teeth supporting removable prosthesis.
* Periapical Abscess or Fistula.
* Patients with systemic disease.
* Patients with xerostomia.
* Participants with a history of allergy to any component of restorations will be used in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
(Marginal adaptation) | 12 months
  (USPHS) criteria

SECONDARY OUTCOMES:
Clinical performance (Anatomical form, Secondary caries, marginal discoloration, Postoperative sensitivity, Color match, Retention) | 12 months
  (USPHS) criteria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Expecting to have all the data by October 2022

REFERENCES:
- [Derived] Al-Salamony H, Akah M, Naguib EA, Safwat OM. Clinical Evaluation of Bulk-fill Alkasite Restoration vs Resin-modified Glass Ionomer in Class V Carious Lesions: 1-year Randomized Clinical Trial. J Contemp Dent Pract. 2024 Dec 1;25(12):1127-1134. doi: 10.5005/jp-journals-10024-3787. PMID 40079991